CLINICAL TRIAL: NCT00139217
Title: NO Need to Ventilate: A Trial of Non-invasive iNO in Persistent Pulmonary Hypertension of the Newborn
Brief Title: NO Need to Ventilate: A Trial of Non-invasive Inhaled Nitric Oxide in Persistent Pulmonary Hypertension of the Newborn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, William T. Mahle, MD, Associate Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1386-2004
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Pulmonary Hypertension
Keywords: Persistent pulmonary hypertension; Non-invasive inhaled nitric oxide; iNO
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: iNO
Procedure: Non-invasive nitric oxide

SUMMARY:
The primary objective of the trial is to determine the feasibility and clinical safety and efficacy of non-invasive inhaled nitric oxide in infants with PPHN without significant pulmonary +-parenchymal disease who would normally receive inhaled nitric oxide only after placement of a tracheal tube and the institution of mechanical ventilation.

DETAILED DESCRIPTION:
Blending low doses of NO gas with oxygen in the inspiratory limb of mechanical ventilators is an effective method for reducing pulmonary vascular resistance and decreasing extrapulmonary right-to-left shunting at the ductus arteriosus and foramen ovale in many patients with PPHN. However, in some patients with PPHN, sustained elevations of PVR may occur in the absence of or despite improvement in the parenchymal lung disease such that mechanical ventilation is not needed for maintaining adequate gas exchange.

PPN in the absence of pulmonary parenchymal disease or despite improvement in the parenchymal lung disease occurs in a significant subset of newborn infants with hypoxemic respiratory failure. Inhaled NO can be effectively delivered by non-invasive techniques to newborn infants with PPHN, potentially reducing the duration of mechanical ventilation, while safely treating the elevation in pulmonary artery pressure and right-to-left.

A dose of 10-20 ppm measured within the delivery device is sufficient to maintain nasopharyngeal concentrations within a range of 1-10 ppm. My co-authors and I have also reported a series of eleven infants with pulmonary hypertension treated with low dose iNO delivered via nasal cannula after extubation at the 14th Annual CNMC Symposium on ECMO & Advanced Therapies for Respiratory Failure, Keystone, CO, 1998.

ELIGIBILITY:
Inclusion Criteria:

* Newborn infants >/= 34 weeks with clinical or echocardiographic evidence of PPHN with a PaO2 < 100 of Fio2 0.8 who are not mechanically ventilated

Exclusion Criteria:

* Infants with significant lung disease
* Inability to sustain spontaneous respirations
* Lethal congenital anomalies
* Severe birth asphyxia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-08; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
% subjects assigned to non-invasive iNO who do not require intubation and mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Golde Dudell, M.D., Principal Investigator — Emory University, Department of Pediatrics, Division of Neonatology
Locations (1):
- Emory University affiliated newborn intensive care units, Atlanta, Georgia, United States